CLINICAL TRIAL: NCT05521724
Title: The Effect of Exercise Training on Individuals With Osteoporotic Vertebral Fractures
Brief Title: Osteoporotic Vertebral Fractures and Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Yasemin Salkin, LECTURER, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HasanKU-YASEMİNSALKİN-1992
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Exercise Addiction; Vertebral Fracture
Keywords: exercise; geriatrics; vertebral fracture; pain
MeSH Terms: conditions — Spinal Fractures; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): The exercise protocol includes balance training and resistance training for all major muscle groups. The program will be performed twice a week.
  * Squat
  * Step up
  * Step-up sideways
  * Upright row
  * Chest presS
  * Biceps curl In balance exercises; It will start with static balance exercises and progress to dynamic balance exercises and will be applied 2 days a week for a minimum of 15 minutes.
  * Tandem stance
  * Semitandem stance
  * Standing exercises on one leg will be performed first with eyes open and then with eyes closed.
  As dynamic balance exercises;
  * Just tip toe walking
  * Don't just walk on heels
  * Tandem walking is selected.
  Interventions: Procedure: exercise
- control group (Active Comparator): No intervention will be made to the control group during the study.
  Interventions: Procedure: exercise

INTERVENTIONS:
Procedure: exercise — resistance and strengthening exercises will be applied to a randomized patient group.

SUMMARY:
Physiotherapy has an important place in the treatment of osteoporotic vertebral fractures. Therapeutic exercise is often recommended for patients with vertebral fractures to reduce pain and restore functional movement. There is not enough evidence in the literature to determine the effects of long-term exercise on osteoporotic fractures and their side effects.

Therefore, the aim of this study is to evaluate the effectiveness of 12-week exercise training in patients with osteoporotic vertebral fractures.

DETAILED DESCRIPTION:
Osteoporotic vertebral fractures are associated with increased morbidity (eg, pain, poor quality of life) and mortality. Therapeutic exercise is a conservative non-pharmacological treatment that is often recommended for patients with vertebral fractures to reduce pain and restore functional movement.

There are preliminary studies showing that exercise may have an important role in improving quality of life and reducing the risk of re-fracture in these individuals. There are several reports of pain relief after short-term (6-10 weeks) exercise programs in people with spinal fractures, suggesting that there is uncertainty in the effects reported after longer-term (12-24 weeks) exercise. Data are scarce and there are only four studies examining this question, and one is a multi-component physical therapy intervention that includes exercise. Not all studies have examined individuals with severe pain at baseline. The quality assessment of the evidence for the effects of exercise on pain is very low.

There is insufficient evidence in the literature to determine the effects of exercise on osteoporotic fractures and their side effects.

Therefore, the aim of the study is to evaluate the effectiveness of 12-week resistance and balance exercises in patients with osteoporotic vertebral fractures.The group of patients who will exercise will be compared with individuals who do not receive any treatment or exercise.

It is aimed to reveal the effects of exercise on pain, physical performance, quality of life, depression, loss of function, kinesiophobia and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory,
* 55 years and over,
* A minimum pain score of 3 in the Short Form Mc-Gill, which we will use for pain assessment.
* Able to use mobile phone by himself or with the support of his family,
* Having at least one vertebral fracture at least 6 months ago as a result of X-ray,
* It was defined as having osteoporosis (Lumbar spine DEXA T score <-2.5).

Exclusion Criteria:

* Metabolic disease that will prevent participation in exercise,
* Pain at a level that prevents participation in exercise (a score above 7 in Short Form Mc Gill)
* Severe cardiovascular or pulmonary diseases (such as Uncontrolled Hypertension, resting heart rate 100 beats/min),
* Psychiatric diseases
* Determined as a recent fracture history

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | A day before the treatment
  The assessment of low back pain will be performed with the Short Form McGill Pain Scale. The form consists of three parts. In the first part, there are 15 descriptive word groups. Of these, 11 evaluate the sensory dimension of the pain, and 4 evaluate the perceptual dimension. These descriptors are rated on an intensity scale from 0 to 3 (0= none, 1= Mild, 2=Moderate, 3= Excess). In the first part of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score and total pain score. In the second part of the form, there are five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. In the third part, the current pain intensity of the patient is evaluated using a visual comparison scale.
Pain Assessment | within 1 week of study completion (average 12 weeks)
  The assessment of low back pain will be performed with the Short Form McGill Pain Scale. The form consists of three parts. In the first part, there are 15 descriptive word groups. Of these, 11 evaluate the sensory dimension of the pain, and 4 evaluate the perceptual dimension. These descriptors are rated on an intensity scale from 0 to 3 (0= none, 1= Mild, 2=Moderate, 3= Excess). In the first part of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score and total pain score. In the second part of the form, there are five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. In the third part, the current pain intensity of the patient is evaluated using a visual comparison scale.

SECONDARY OUTCOMES:
Physical Performance Assessment | within 1 week of study completion (average 12 weeks)
  A 6 Minute Walk Test will be used. It is a functional walking capacity test in which patients walk at their own pace. Patients walk as far as they can in a straight corridor in six minutes. Standardized commands and words of encouragement are used. Primary endpoint: Six-minute walk.
Quality of Life Assessment | within 1 week of study completion (average 12 weeks)
  The European Osteoporosis Foundation Quality of Life Questionnaire-41 will be used to assess patients' quality of life.
  The European Osteoporosis Foundation Quality of Life Questionnaire-41, such as pain (5 items), physical function (17 items), social activity (7 items), general health assessment (3 items) and mental function (9 items); It consists of 5 subscales that examine the five dimensions of health. The answers to the questions in the QUALEFFO-41 scale are scored from 1 (healthy) to 5 (unhealthy), respectively. The section score and the total score are calculated by transferring the scores to a measurement out of 100. For each subgroup and overall outcome in the scale, 0 points indicate the best health status, while 100 points indicate the worst health status.
Depression Assessment | within 1 week of study completion (average 12 weeks)
  Beck Depression Scale will be used to evaluate the depression of the patients. The Beck Depression Scale consists of 21 questions questioning behavior and feelings related to the general depressive state. A high score indicates increased depressive symptom severity. It was developed to measure the risk of depression, the level of depressive symptoms and the change in severity in adults. Turkish validity and reliability study was done by Hisli. It contains a total of 21 self-evaluation sentences. Each item receives an increasing score between 0-3 and the total varies between 0-63. In the validity and reliability article of the scale for Turkish, the cut-off point was accepted as 17. Scores of eighteen and above are considered to be indicative of moderate and severe depression.
Loss of Function Assessment | within 1 week of study completion (average 12 weeks)
  The Oswestry Disability Index will be used to assess the degree of loss of function due to low back pain. The Turkish validity and reliability of the Oswestry Disability Index, which was demonstrated in 2004, consists of 10 items. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, the degree of change in pain, travel and social life. Under each item, there are six statements that the patient marked as appropriate for his/her condition. The first statement is scored as "0" and the sixth statement is scored as "5". When the total score is calculated, it is multiplied by two and expressed as a percentage. The maximum score is "100", the minimum score is "0". As the total score increases, the level of disability also increases.
Kinesiophobia Assessment | within 1 week of study completion (average 12 weeks)
  The Tampa Kinesiophobia Scale, which is based on the fear of avoidance due to fear constituting pain-based movement limitation, fear in work-related activities, fear of movement or re-injury, and the Turkish version of the scale and the reliability study of the scale, will be used in the assessment of kinesiophobia. The Tampa kinesiophobia scale is a 17-item scale developed to measure the fear of movement or re-injury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. A 4-point Likert scoring (1=strongly disagree, 4=strongly agree) is used in the scale. After reversing items 4, 8, 12 and 16, a total score is calculated. In this evaluation, the individual gets a score between 17-68. A high score on the scale indicates that kinesiophobia is also high.
Sleep Quality Assessment | within 1 week of study completion (average 12 weeks)
  It will be evaluated by the Pittsburgh Sleep Quality Index. The Pittsburgh Sleep Quality Index is a 19-item self-report scale that assesses sleep quality and impairment over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are questions to be answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleeping Drug Use, and Daytime Dysfunction. Each component is evaluated over 0-3 points. The total score of the 7 components gives the scale total score. The total score ranges from 0 to 21. A total score greater than 5 indicates "poor sleep quality"
Sleepiness State Assessment | within 1 week of study completion (average 12 weeks)
  Sleepiness will be evaluated with the Epworth Sleepiness Scale. It is a simple, easy-to-understand, 8-item scale with proven validity and reliability in assessing the general sleepiness level in adults. In the survey, participants are asked to evaluate the probability of falling asleep during the activities they do during the day, although not every day, and evaluate them on a scale of 0 to 3. The questionnaire consists of a total of 8 situations. While the score between 0-9 obtained as a result of the survey is considered as normal, the score between 10-24 indicates that the expert should be consulted. Scores between 11 and 15 indicate mild to moderate sleep apnea, while scores of 16 and above indicate severe sleep apnea or narcolepsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin Üniversitesi, Mersin, Yeni̇şehi̇r/mersi̇n, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbs JC, MacIntyre NJ, Ponzano M, Templeton JA, Thabane L, Papaioannou A, Giangregorio LM. Exercise for improving outcomes after osteoporotic vertebral fracture. Cochrane Database Syst Rev. 2019 Jul 5;7(7):CD008618. doi: 10.1002/14651858.CD008618.pub3. PMID 31273764
- [Background] Barker KL, Newman M, Stallard N, Leal J, Minns Lowe C, Javaid MK, Noufaily A, Adhikari A, Hughes T, Smith DJ, Gandhi V, Cooper C, Lamb SE. Exercise or manual physiotherapy compared with a single session of physiotherapy for osteoporotic vertebral fracture: three-arm PROVE RCT. Health Technol Assess. 2019 Aug;23(44):1-318. doi: 10.3310/hta23440. PMID 31456562
- [Result] Giangregorio LM, Papaioannou A, Macintyre NJ, Ashe MC, Heinonen A, Shipp K, Wark J, McGill S, Keller H, Jain R, Laprade J, Cheung AM. Too Fit To Fracture: exercise recommendations for individuals with osteoporosis or osteoporotic vertebral fracture. Osteoporos Int. 2014 Mar;25(3):821-35. doi: 10.1007/s00198-013-2523-2. Epub 2013 Nov 27. PMID 24281053
- See also: ARTICLE 1 — http://pubmed.ncbi.nlm.nih.gov/31456562/
- See also: ARTICLE 2 — http://pubmed.ncbi.nlm.nih.gov/31273764/
- See also: ARTICLE 3 — http://pubmed.ncbi.nlm.nih.gov/24281053/